CLINICAL TRIAL: NCT05532514
Title: EFFECT OF LIMITED VOLUME CONE BEAM COMPUTED TOMOGRAPHY ON MICRONUCLEI CELLS COUNT OF BUCCAL MUCOSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Dr.Komal Kumia
Record Dates: First submitted 2022-09-03; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Micronuclei Count

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Buccal epithelial cells will be collected from each subject by principal investigator which will be subjected to exfoliative cytology. Prior to cell collection, the patients will be asked to rinse their mouth with water to remove saliva, food particles or any other debris. Cells will be obtained by gentle scraping with a metal spatula and transferred to a tube containing normal saline which will be followed by centrifugation at the rate of 1000rpm for 3 min, thrice. The suspension will be fixed with a fixative (methanol: acetic acid in the ratio 3:1) dropped onto the clean slides after that slides to be stained by the Papanicolaou stain.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP A: exposure in 5x5 fov at 90 voxel size
  Interventions: Other: MICRONUCLEI COUNT
- GROUP B: exposure in 5x5 fov at 200 voxel size
  Interventions: Other: MICRONUCLEI COUNT

INTERVENTIONS:
Other: MICRONUCLEI COUNT — MICRONUCLEI COUNT IN PRECBCT and POSTCBCT EXPOSURE

SUMMARY:
title -Effect of limited Cone Beam Computed Tomography on micronucleated cell count of buccal mucosa.

Rationale: Our study aims to detect and establish a correlation between mean micronucleated cell count and nuclear morphometry in exfoliated cells from affected and apparently unaffected mucosa after CBCT radiation and compare them with exfoliated cells from normal appearing mucosa of normal subjects before CBCT. This could prove beneficial in early detection of malignant conversion of buccal mucosa after CBCT and hence improve the prognosis and better treatment outcome of the patient.

RESEARCH QUESTION-what is the effect of CBCT radiations on the no. Of micronucleated cells in the buccal mucosal cells Population- Patients Planned For CBCT Intervention- None Control-None Outcome- change in number of mean micronucleated cell count before and after the CBCT exposure Time- 1 year (Jan 2020- April 2021)

DETAILED DESCRIPTION:
Ionizing radiation is a well-known mutagen and carcinogen in the human population which has both direct and indirect effects on the tissues. It can damage the tissues through different mechanisms like breakage, cross linking of DNA strands, change or loss of the base and disruption of hydrogen bonds. These radiations cause changes in the buccal mucosa, salivary glands, dentin and enamel leading to xerostomia, mucositis and radiation related caries.

Buccal mucosal cells are under direct radiation exposure in dental radiographic techniques and act as the primary target for radiation-induced damage. Also, it has a highly proliferative epithelial cells and can be easily collected and studied. Micronuclei, an anomaly structure, originates from the chromosome fragments or whole chromosomes that lag behind at anaphase during nuclear division under physical and chemical factors. The micronucleus index has become one of the standard cytogenetic endpoints and biomarkers used in genetic toxicology in vivo or in vitro2. In healthy epithelial tissues these MNi ranges from 0.5 to 2.5 MNi /1000 cells. The studies have shown an increase in their frequency in individuals exposed to radiation or other genotoxic agents.

However, these studies observed the effect on the micronuclei at small and medium FOV, but the radiation induced damage is seen mostly at smaller FOVs which involves high resolution, thereby causing more radiation exposure.

Keeping this in mind, the aim of this study is to observe and correlate the mean micro nucleated cell count of the buccal epithelial cells with the help of PAP smear after CBCT exposure at different voxel sizes (90 and 200) at small FOV. This could prove beneficial and shed light on the cytogenetic damage and malignant conversion potential of buccal mucosa after CBCT.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals

Exclusion Criteria:

- Subjects with any other potentially malignant disorder present in the oral cavity. .

2. Subjects who are smokers and alcoholics. 3. Subjects with history of malignancy. 4. Subjects receiving dietary supplementations 5. Any subjects exposed to radiation or other carcinogens in the past one month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - patient reporting to oral radiology for CBCT for any dental conditions
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
THE CHANGE IN NUCLEAR DIMENSIONS WILL BE NOTICED AFTER CBCT EXPOSURE | 1 YEAR
  MICROSCOPIC ANALYSIS WITH PAP SMEAR OF EXFOLIATED CELLS

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute Of Dental Science, Rohtak, Haryana, India

REFERENCES:
- [Background] Arora P, Devi P, Wazir SS. Evaluation of genotoxicity in patients subjected to panoramic radiography by micronucleus assay on epithelial cells of the oral mucosa. J Dent (Tehran). 2014 Jan;11(1):47-55. Epub 2014 Jan 31. PMID 24910676
- [Background] Thomas P, Holland N, Bolognesi C, Kirsch-Volders M, Bonassi S, Zeiger E, Knasmueller S, Fenech M. Buccal micronucleus cytome assay. Nat Protoc. 2009;4(6):825-37. doi: 10.1038/nprot.2009.53. Epub 2009 May 7. PMID 19444240
- [Background] da Fonte JB, Andrade TM, Albuquerque RL Jr, de Melo MFB, Takeshita WM. Evidence of genotoxicity and cytotoxicity of X-rays in the oral mucosa epithelium of adults subjected to cone beam CT. Dentomaxillofac Radiol. 2018 Feb;47(2):20170160. doi: 10.1259/dmfr.20170160. Epub 2017 Nov 13. PMID 29091472
- [Background] Popova L, Kishkilova D, Hadjidekova VB, Hristova RP, Atanasova P, Hadjidekova VV, Ziya D, Hadjidekov VG. Micronucleus test in buccal epithelium cells from patients subjected to panoramic radiography. Dentomaxillofac Radiol. 2007 Mar;36(3):168-71. doi: 10.1259/dmfr/29193561. PMID 17463102
- [Background] Belmans N, Gilles L, Virag P, Hedesiu M, Salmon B, Baatout S, Lucas S, Jacobs R, Lambrichts I, Moreels M. Method validation to assess in vivo cellular and subcellular changes in buccal mucosa cells and saliva following CBCT examinations. Dentomaxillofac Radiol. 2019 Sep;48(6):20180428. doi: 10.1259/dmfr.20180428. Epub 2019 Apr 5. PMID 30912976
- [Background] Antonio EL, Nascimento AJD, Lima AAS, Leonart MSS, Fernandes A. GENOTOXICITY AND CYTOTOXICITY OF X-RAYS IN CHILDREN EXPOSED TO PANORAMIC RADIOGRAPHY. Rev Paul Pediatr. 2017 Jul-Sep;35(3):296-301. doi: 10.1590/1984-0462/;2017;35;3;00010. Epub 2017 Jul 20. PMID 28977295